CLINICAL TRIAL: NCT03256123
Title: The Effect of Biscuits Containing Red Palm Oil on School Children With Vitamin A Deficiency in West and East Malaysia
Brief Title: The Effects of Biscuits Containing Red Palm Oil on School Children With Vitamin A Deficiency in West and East Malaysia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD219/16
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-11

CONDITIONS: Vitamin A Deficiency in Children
Keywords: Vitamin A Deficiency; Iron Deficiency; Parasite; Gut Microbiota; Red palm oil
MeSH Terms: conditions — Vitamin A Deficiency; Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: In this study, the subjects will be randomly assigned to two groups: a group receiving biscuits with red palm olein shortening and a control group receiving biscuits with palm olein shortening with corresponding fatty acids.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- red palm shortening group (Experimental): A group receiving the supplementation of red palm shortening biscuits. The subjects are expected to receive 326.3 µg RE of vitamin A/day by consuming the biscuits four days a week.
  Interventions: Dietary Supplement: red palm shortening group
- palm shortening group (Placebo Comparator): A group receiving supplementation of palm shortening biscuits with corresponding fatty acids as red palm shortening group.
  Interventions: Dietary Supplement: palm shortening group

INTERVENTIONS:
Dietary Supplement: red palm shortening group — Biscuits made of red palm shortening will be distributed to the subjects given four days a week on schooling days for a duration of 6 months. This biscuit would be given four days a week on schooling days for a duration of 6 months. On average in a week, subject is expected to receive 326.3 µg RE of vitamin A/day. This would fulfill ~59.3% of the RNI of vitamin A for children aged 7-12 years old.
  Arms: red palm shortening group
Dietary Supplement: palm shortening group — Biscuits made of palm shortening (control group) will be distributed to the subjects given four days a week on schooling days for a duration of 6 months. The palm shortening biscuits contain corresponding fatty acids as red palm shortening group.
  Arms: palm shortening group

SUMMARY:
Based on recent nutrition survey (SEANUTS Malaysia) on a total of 3542 Malaysian Children aged between 6 months to 12 years old, 4.4% of the children had vitamin A deficiency. Rural areas recorded a higher prevalence of vitamin A deficiency (6.4%) compared with urban areas (3.8%). Besides, prevalence of iron deficiency due to low ferritin concentrations is 4.4% and anaemia based on low haemoglobin concentrations is 6.6%. It is proposed that a red palm oil intervention programme to be conducted in alliance with RMT in Malaysia to enhance the Vitamin A status of school children in underprivileged community in Malaysia.

DETAILED DESCRIPTION:
Deficiency of vitamin A or retinol is a public health problem and listed as the most widespread nutritional deficiency worldwide (Sommer, 1995). According to the World Health Organization (WHO), about 190 million preschool children in underdeveloped countries especially in the region of Africa and South-East Asia are vitamin A deficient (2011, 2011). Infants and children have higher vitamin A requirements to promote rapid growth and better immunity to combat infections. Vitamin A deficiency in children causes visual impairment and blindness, risk of infection, stunting, anemia, respiratory diseases and mortality due to common childhood infections such as diarrhea and measles. On the basis on Cochrane meta-analysis on 194,795 children, vitamin A supplementation could reduce childhood mortality by 23% and incidences of illnesses (Imdad et al., 2010).

According to WHO, an estimated 2.8 million preschool-age children are at risk of nutritional blindness or active xerophthalmia due to Vitamin A deficiency in low-income countries (Organization, 2010). Sadly, approximately 250 000 to 500 000 children suffering from vitamin A deficiency become blind yearly, and half of the number die within a year of losing their vision (Organization, 2010). The different eye signs of vitamin A deficiency (VAD) in children as graded by the WHO are night blindness, conjunctival xerosis, Bitot's spots, corneal xerosis, corneal ulcer/keratomalacia and corneal scarring (Sommer, 1995). Severe vitamin A deficiency distresses ocular tissue by reducing regeneration of visual pigment upon exposure to bright light or lasting damage on the epithelium of the cornea and conjunctiva. Classical ocular manifestation due to vitamin A deficiency may lead to less serious Bitot's spots and night blindness, or severe xerophthalmia and keratomalacia leading to blindness (Scrimshaw, 2000). Ocular manifestation of vitamin A deficiency still exists in underprivileged communities in Malaysia (Ngah et al., 2002). Vitamin A deficiency is prevalent in pre-school and primary school children of aborigines ("Orang Asli") and those from rubber estates. 82.2% of Orang Asli children had ocular manifestations of vitamin A deficiency ranging from history of night blindness to corneal scars (Ngah et al., 2002). Based on recent nutrition survey (SEANUTS Malaysia) on a total of 3542 Malaysian Children aged between 6 months to 12 years old, 4.4% of the children had vitamin A deficiency. Rural areas recorded a higher prevalence of vitamin A deficiency (6.4%) compared with urban areas (3.8%) (Poh et al., 2013).

There is significant association between iron deficiency and vitamin A deficiency represented by low serum retinol (Al-Mekhlafi et al., 2013). According to WHO, iron deficiency is the commonest and widespread nutritional deficiency in the world. Over 30% of the world's population are known to be anaemic due to iron deficiency, poor diet, or exposed to infectious diseases. Malaria, HIV/AIDS, hookworm infestation, schistosomiasis, and other infections such as tuberculosis are particularly important factors contributing to the high prevalence of anaemia in some areas. Iron deficiency may lead to impaired health, development and learning in children. Based on Malaysian SEANUTS survey, the overall prevalence of iron deficiency due to low ferritin concentrations is 4.4% and anaemia based on low haemoglobin concentrations is 6.6% (Poh et al., 2013). The occurrence of anaemia and iron deficiency among Orang Asli children is relatively high. The Orang Asli children aged 2-15 years old, living in eight villages in Selangor showed high episodes of anaemia 41.5% and 36.5% had iron deficiency anaemia. In another recent study, nearly half (48.5%) of the Orang Asli children from 18 villages in Pahang were found to be anaemic and the prevalence of iron deficiency was 34% (Al-Mekhlafi et al., 2013).

In Malaysia, the school-feeding program is called "Rancangan Makanan Tambahan (RMT)" which literally means additional food plan. The RMT program is provided only to primary school children (aged 6 - 12 years) from poor families. It is not meant to replace food served at home, but to provide extra nourishment for children from poor families. The RMT program is managed by the School Division of the Ministry of Education, Malaysia. Food is served during recess time (10.30 a.m. for morning session, and 3.30pm for afternoon session) and provides 1/4 to 1/3 of daily requirements. It is proposed that a red palm oil intervention programme to be conducted in alliance with RMT in Malaysia to enhance the Vitamin A status of school children in underprivileged community in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-11 years old
* Vitamin A deficient children defined as concentration of serum retinol <0.70 µmol/L and suspected vitamin A deficiency defined as concentration of serum retinol 0.70 - <1.05 µmol/L.
* Not physically handicapped

Exclusion Criteria:

* Children with oedema including severe acute malnutrition or gastrointestinal disorders
* Children allergic to wheat- and/or gluten-containing foods
* Children who are studying Primary Six

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 651 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Retinol level | During screening, after 6 months of dietary intervention period and post 200 days after the intervention.
  Vitamin A deficiency is defined as concentration of blood retinol <0.70 µmol/L and suspected vitamin A deficiency is defined as concentration of blood retinol 0.70 - <1.05 µmol/L.

SECONDARY OUTCOMES:
Plasma beta carotene, alpha carotene, vitamin E levels | at the baseline, after 6 months of dietary intervention period and post 200 days after the intervention.
  Plasma beta carotene, alpha carotene, vitamin E levels are lower in Vitamin A deficiency kids
Retinol binding protein levels | at the baseline, after 6 months of dietary intervention period and post 200 days after the intervention.
  Retinol is transported in a 1-to-1 complex with retinol-binding protein. The cutoff of equimolar RBP is able to predict vitamin A deficiency
Haematological markers | at the baseline, after 6 months of dietary intervention period and post 200 days after the intervention.
  vitamin A is essential for normal haematopoiesis. The occurrence of anaemia is indicated by haemoglobin concentration lower than 115 g/L. The occurrence of iron deficiency is indicated by the serum ferritin concentration lower than 15 μg/L.
Ocular signs | at the baseline, after 6 months of dietary intervention period and post 200 days after the intervention.
  Eyes examined at optimal light for conjuctival xerosis, Bitot's spots, corneal xerosis, and corneal ulceration or keratomalacia. The eye assessments include visual acuity assessment via a Snellen chart, examination with a portable slit lamp for signs of xerophthalmia, fundus photography with portable non mydriatic camera and questionnaire on night blindness symptoms.
Inflammatory/infection status | at the baseline, after 6 months of dietary intervention period and post 200 days after the intervention.
  high sensitivity C-reactive protein (hsCRP), haematology tests
Gut Microbiota | at the baseline, 3 months after intervention and after 6 months of dietary intervention period.
  As malnutrition is generally associated with the changes in gut microbiota [14], it is important to study the effects of red palm oil-fortified biscuit supplementation to gut microbiota of VAD children.
Soil-transmitted helminth | at the baseline, 3 months after intervention and after 6 months of dietary intervention period.
  Malnutrition can weaken immune responses and increase the susceptibility to parasitic infections. Therefore, the supplementation of vitamin A to VAD children has the potential to boost their immunity against parasitic reinfections.

CONTACTS AND LOCATIONS:
Overall Officials: KIM TIU TENG, Principal Investigator — Malaysia Palm Oil Board; RADHIKA LOGANATHAN, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gemmell HG, Smith FW, Innes A, Edward N, Catto GR. The value of Tc-DTPA transit times and NMR T1 measurements in monitoring the progress of renal transplants. Nucl Med Commun. 1985 Feb;6(2):67-74. PMID 3916855
- [Background] van Stuijvenberg ME, Faber M, Dhansay MA, Lombard CJ, Vorster N, Benade AJ. Red palm oil as a source of beta-carotene in a school biscuit used to address vitamin A deficiency in primary school children. Int J Food Sci Nutr. 2000;51 Suppl:S43-50. doi: 10.1080/096374800750049567. PMID 11271856
- [Background] Zeba AN, Martin Prevel Y, Some IT, Delisle HF. The positive impact of red palm oil in school meals on vitamin A status: study in Burkina Faso. Nutr J. 2006 Jul 17;5:17. doi: 10.1186/1475-2891-5-17. PMID 16846498
- [Derived] Tan PY, Lim CC, Seng KBH, Loganathan R, Lim YA, Teng KT, Mohd Johari SN, Selvaduray KR, Ramli N. Red palm olein supplementation as a potential preventive solution for xerophthalmia among vitamin A-deficient primary schoolchildren: a cluster randomized controlled trial. Eur J Clin Nutr. 2025 Sep;79(9):928-936. doi: 10.1038/s41430-025-01620-2. Epub 2025 Apr 17. PMID 40247111
- [Derived] Tan PY, Loganathan R, Teng KT, Mohd Johari SN, Lee SC, Selvaduray KR, Ngui R, Lim YA. Supplementation of red palm olein-enriched biscuits improves levels of provitamin A carotenes, iron, and erythropoiesis in vitamin A-deficient primary schoolchildren: a double-blinded randomised controlled trial. Eur J Nutr. 2024 Apr;63(3):905-918. doi: 10.1007/s00394-023-03314-6. Epub 2024 Jan 19. PMID 38240773